CLINICAL TRIAL: NCT02916407
Title: The Effect of Preoperative Ketamine on the Emergence Characteristics After Desflurane or Sevoflurane Anesthesia in Children Undergoing Entropion Surgery
Brief Title: The Effect of Preoperative Ketamine on the Emergence Characteristics in Children Undergoing Entropion Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Ki Hwa Lee, Assistant professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2016-01
Record Dates: First submitted 2016-09-01; First posted 2016-09-27 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Entropion
Keywords: Anesthesia; Agitation; Extubation
MeSH Terms: conditions — Entropion; Psychomotor Agitation | interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane Group (Active Comparator): The patients will maintained general anesthesia with sevoflurane.
  Interventions: Drug: Sevoflurane
- Desflurane Group (Experimental): The patients will maintained general anesthesia with desflurane.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — Intravenous ketamine will administrate to the patients for decreasing of separation anxiety of children.
  General anesthesia will maintained with sevoflurane 2-3 vol%.
  Other Names: sevofrane
  Arms: Sevoflurane Group
Drug: Desflurane — Intravenous ketamine will administrate to the patients for decreasing of separation anxiety of children.
  General anesthesia will maintained with desflurane 6-7vol%.
  Other Names: suprane
  Arms: Desflurane Group

SUMMARY:
The investigators evaluate extubation time and recovery profiles in children undergoing entropion surgery.

DETAILED DESCRIPTION:
This study will compare the extubation time and recovery profiles (degree of postoperative agitation and cough) between sevoflurane group and desflurane group. General anesthesia will maintained with sevoflurane 2-3vol% or desflurane 6-7vol%. After surgery, the investigators will measure the duration of extubation and recovery profiles between two groups.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologist class 1 patients
* 3-6 years children undergoing entropion surgery

Exclusion Criteria:

* Do not agree with participate this study

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2016-09; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ki Hwa Lee, M.D,, Principal Investigator — Inje University
Locations (1):
- Haeundae paik hospital, inje university, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 56 patients were enrolled in this study and no patient was dropped.
Groups:
- Sevoflurane Group: The patients will maintained general anesthesia with sevoflurane.
  Sevoflurane: Intravenous ketamine will administrate to the patients for decreasing of separation anxiety of children.
  General anesthesia will maintained with sevoflurane 2-3 vol%.
- Desflurane Group: The patients will maintained general anesthesia with desflurane.
  Desflurane: Intravenous ketamine will administrate to the patients for decreasing of separation anxiety of children.
  General anesthesia will maintained with desflurane 6-7vol%.
Period: Overall Study
Arm/Group | Sevoflurane Group | Desflurane Group
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 56 patients were enrolled in this study and no patient was dropped.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sevoflurane Group | Desflurane Group | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.3 (1.1) | 4.6 (1.1) | 4.5 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 15 | 14 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 28 | 28 | 56
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 28 | 28 | 56
Height [Mean (Standard Deviation); unit: centimeter] — centimeter
  centimeter | 107.8 (7.4) | 108.6 (9.9) | 108.2 (8.722)

OUTCOME MEASURES:

1. Primary Outcome: Extubation Time
Description: compare the extubation time between sevoflurane and desflurane group
Time Frame: 30 minutes
Population: A total of 56 patients were enrolled in this study and no patient was dropped.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sevoflurane Group | Desflurane Group
Number analyzed (Participants) | 28 | 28
seconds | 756.3 (267.2) | 425.9 (122.9)

2. Secondary Outcome: Degree of Postoperative Agitation
Description: Postoperative agitation will measure using Pediatric Anesthesia Emergence Delirium (PAED) scale. PAED scale is "(1) The child makes eye contact with the caregiver (2) The child's action are purposeful (3) The child is aware of his/her surrounding (4) The child is restless (5) The child is inconsolable." It scores 0-4, and total maximum score is 20.
  PAED score > 12 was used to determine occurence of postoperative agitation.
Time Frame: 30 minutes
Population: A total of 56 patients were enrolled in this study and no patient was dropped.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Sevoflurane Group | Desflurane Group
Number analyzed (Participants) | 28 | 28
units on a scale | 15 [6 to 20] | 10 [5 to 20]

ADVERSE EVENTS:
Time Frame: 30 minutes after surgery
Description: There was no serious adverse event.
Arm/Group | Sevoflurane Group | Desflurane Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 5/28 | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sevoflurane Group (N=28) | Desflurane Group (N=28)
copious secretion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
desaturation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
There was non-ketamine (control) group. We used ketamine for reducing of separation anxiety of children.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT02916407/Prot_SAP_000.pdf